CLINICAL TRIAL: NCT05738486
Title: Investigating the Effect of Different Donanemab Dosing Regimens on ARIA-E and Amyloid Lowering in Adults With Early Symptomatic Alzheimer's Disease
Brief Title: A Study of Different Donanemab (LY3002813) Dosing Regimens in Adults With Early Alzheimer's Disease (TRAILBLAZER-ALZ 6)
Status: Active, not recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Eli Lilly and Company (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 18648; I5T-MC-AACQ (Other: Eli Lilly and Company); 2022-502268-18-00 (Other: EU Trial Number); U1111-1285-9438 (Other: UTN Number)
Record Dates: First submitted 2023-02-13; First posted 2023-02-22 (Actual); Results first posted 2025-11-14 (Actual); Last update posted 2025-11-14 (Actual); Status verified 2025-10

CONDITIONS: Alzheimer's Disease; Dementia; Brain Diseases; Central Nervous System Diseases; Nervous System Diseases; Neurodegenerative Diseases; Neurocognitive Disorders; Mental Disorders
MeSH Terms: conditions — Alzheimer Disease; Dementia; Brain Diseases; Central Nervous System Diseases; Nervous System Diseases; Neurodegenerative Diseases; Neurocognitive Disorders; Mental Disorders | interventions — donanemab; Dexamethasone

STUDY DESIGN:
Intervention Model Description: Phase 3b
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (6):
- 1400 mg Donanemab - Standard Regimen (Experimental): Participants received:
  * 700 milligrams (mg) donanemab administered intravenously (IV) at baseline, week 4, and 8.
  * placebo administered IV at week 2, 6, 10, and 14.
  * 1400 mg of donanemab administered IV at week 12, 16, 20, and 24.
  Interventions: Drug: Donanemab; Drug: Placebo
- 1400 mg Donanemab - Dose Skipping (Experimental): Participants received:
  * 700 mg donanemab administered IV at baseline.
  * placebo administered IV at week 2, 4, 6, 10, and 14.
  * 1400 mg of donanemab administered IV at week 8, 12, 16, 20, and 24.
  Interventions: Drug: Donanemab; Drug: Placebo
- 1400 mg Donanemab - Titration (Experimental): Participants received:
  * 350 mg donanemab administered IV at baseline.
  * placebo administered IV at week 2, 6, 10, and 14.
  * 700 mg donanemab administered IV at week 4.
  * 1050 mg of donanemab administered IV at week 8.
  * 1400 mg of donanemab administered IV at week 12, 16, 20, and 24.
  Interventions: Drug: Donanemab; Drug: Placebo
- 1400 mg Donanemab - Maximum Concentration (Cmax) (Experimental): Participants received:
  * 350 mg donanemab administered IV at baseline, weeks 2, 4, 6, 8, and 10.
  * 700 mg donanemab administered IV at weeks 12 and 14.
  * 1400 mg of donanemab administered IV at weeks 16, 20, and 24.
  Interventions: Drug: Donanemab; Drug: Placebo
- Donanemab Addendum Arm 1 (Experimental): Participants will receive donanemab by IV infusion.
  Participants will receive placebo pretreatment to preserve the blind prior to donanemab infusion.
  Interventions: Drug: Donanemab; Drug: Placebo
- Donanemab Addendum Arm 2 (Experimental): Participants will receive donanemab by IV infusion.
  Participants will receive dexamethasone pretreatment prior to donanemab infusion
  Interventions: Drug: Donanemab; Drug: Dexamethasone

INTERVENTIONS:
Drug: Donanemab — Administered IV
  Other Names: LY3002813
Drug: Placebo — Administered IV
  Arms: 1400 mg Donanemab - Dose Skipping; 1400 mg Donanemab - Maximum Concentration (Cmax); 1400 mg Donanemab - Standard Regimen; 1400 mg Donanemab - Titration; Donanemab Addendum Arm 1
Drug: Dexamethasone — Administered IV
  Arms: Donanemab Addendum Arm 2

SUMMARY:
This study will investigate different donanemab dosing regimens and their effect on the frequency and severity of ARIA-E in adults with early symptomatic Alzheimer's disease (AD) and explore participant characteristics that might predict risk of ARIA.

Approximately 375 additional participants will be enrolled per addendum.

The study will last approximately 91 weeks and include up to 26 visits in the main study.

ELIGIBILITY:
Inclusion Criteria:

* Gradual and progressive change in memory function reported by the participant or informant for ≥6 months.
* A mini mental state examination (MMSE) score of 20 to 28 (inclusive) at screening.
* Have an amyloid PET scan result from central read, consistent with the presence of amyloid pathology.

Exclusion Criteria:

* Have significant neurological disease affecting the central nervous system other than AD, that may affect cognition or ability to complete the study, including but not limited to, other dementias, serious infection of the brain, Parkinson's disease, multiple concussions, or epilepsy or recurrent seizures, except febrile childhood seizures.
* Has current serious or unstable illnesses including cardiovascular, hepatic, renal, gastroenterologic, respiratory, endocrinologic, neurologic (other than AD), psychiatric, immunologic, or hematologic disease and other conditions that, in the investigator's opinion, could interfere with the analyses in this study.
* A life expectancy of <24 months.
* Contraindication to MRI or PET scans
* Have had prior treatment with a passive anti-amyloid immunotherapy.
* Have a presence or history of malignant neoplasms within the past 5 years prior to Visit 1.

Exceptions:

* non-metastatic basal- or squamous-cell skin cancer
* Stage 0 non-invasive carcinoma of the cervix
* Stage 0 non-invasive prostate cancer, or
* other cancers with low risk of recurrence or spread

Ages: 60 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1175 (Actual)
Dates: Start 2023-02-28 (Actual); Primary Completion 2024-05-16 (Actual); Study Completion 2027-05 (Estimated)

CONTACTS AND LOCATIONS:
Overall Officials: Call 1-877-CTLILLY (1-877-285-4559) or 1-317-615-4559 Mon - Fri 9 AM - 5 PM Eastern time (UTC/GMT - 5 hours, EST), Study Director — Eli Lilly and Company
Locations (49):
- United States (43):
  - MD First Research - Chandler, Chandler, Arizona
  - Irvine Clinical Research, Irvine, California
  - Healthy Brain Clinic, Long Beach, California
  - California Neuroscience Research Medical Group, Inc., Sherman Oaks, California
  - JEM Research Institute, Atlantis, Florida
  - VIN-Julie Schwartzbard, Aventura, Florida
  - Excel Medical Clinical Trials, Boca Raton, Florida
  - K2 Medical Research, Clermont, Florida
  - Brain Matters Research, Delray Beach, Florida
  - Neuropsychiatric Research Center of Southwest Florida, Fort Myers, Florida
  - Finlay Medical Research, Greenacres City, Florida
  - Infinity Clinical Research, LLC, Hollywood, Florida
  - Jacksonville Center for Clinical Research, Jacksonville, Florida
  - ClinCloud - Maitland, Maitland, Florida
  - K2 Medical Research, Maitland, Florida
  - ClinCloud - Viera, Melbourne, Florida
  - Suncoast Clinical Research, Inc., New Port Richey, Florida
  - Renstar Medical Research, Ocala, Florida
  - Charter Research - Winter Park, Orlando, Florida
  - Progressive Medical Research, Port Orange, Florida
  - Alzheimer's Research and Treatment Center, Stuart, Florida
  - K2 Medical Research - Tampa, Tampa, Florida
  - K2 Summit Research, The Villages, Florida
  - Charter Research - Lady Lake, The Villages, Florida
  - Alzheimer's Research and Treatment Center, Wellington, Florida
  - Palm Beach Neurology, West Palm Beach, Florida
  - Conquest Research, Winter Park, Florida
  - Columbus Memory Center, LLC, Columbus, Georgia
  - CenExel iResearch, LLC, Decatur, Georgia
  - Center for Advanced Research & Education, Gainesville, Georgia
  - CenExel iResearch, LLC, Savannah, Georgia
  - MedVadis Research Corporation, Waltham, Massachusetts
  - Adams Clinical, Watertown, Massachusetts
  - QUEST Research Institute, Farmington Hills, Michigan
  - The Cognitive and Research Center of New Jersey, Springfield, New Jersey
  - Butler Hospital, Providence, Rhode Island
  - Neurology Clinic, P.C., Cordova, Tennessee
  - Gadolin Research, Beaumont, Texas
  - Kerwin Medical Center, Dallas, Texas
  - The University of Texas Health Science Center at Houston, Houston, Texas
  - Re:Cognition Health, Fairfax, Virginia
  - Northwest Clinical Research Center, Bellevue, Washington
  - Universal Research Group, Tacoma, Washington
- United Kingdom (6):
  - Re:Cognition Health - Bristol, Bristol, Bristol, City of
  - Re:Cognition Health - Winchester, Winchester, Hampshire
  - Re:Cognition Health - London, London, London, City of
  - Re:Cognition Health Guildford, Guildford, Reading
  - Re:Cognition Health - Birmingham, Birmingham
  - Re:Cognition Health - Plymouth, Plymouth

IPD SHARING:
Plan to Share IPD: Yes
Anonymized individual patient level data will be provided in a secure access environment upon approval of a research proposal and a signed data sharing agreement.
Supporting Information: Study Protocol, SAP, CSR
Time Frame: Data are available 6 months after the primary publication and approval of the indication studied in the US and European Union (EU), whichever is later. Data will be indefinitely available for requesting.
Access Criteria: A research proposal must be approved by an independent review panel and researchers must sign a data sharing agreement.
URL: http://vivli.org/

REFERENCES:
- [Derived] Wang H, Nery ESM, Ardayfio P, Khanna R, Svaldi DO, Shcherbinin S, Xu W, Andersen SW, Hauck PM, Brooks DA, Collins EC, Salloway S, Mintun MA, Sims JR. The effect of modified donanemab titration on amyloid-related imaging abnormalities with edema/effusions and amyloid reduction: 18-month results from TRAILBLAZER-ALZ 6. J Prev Alzheimers Dis. 2025 Sep;12(8):100266. doi: 10.1016/j.tjpad.2025.100266. Epub 2025 Jul 5. PMID 40619285
- See also: A Study of Different Donanemab (LY3002813) Dosing Regimens in Adults With Early Alzheimer's Disease (TRAILBLAZER-ALZ 6) — https://trials.lilly.com/en-US/trial/389475

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Current results reporting is for primary results completion date (16-May-2024) i.e., up to week 24. Data beyond week 24 will be reported at the time of final results reporting.
Pre-assignment Details: Addendum recruited a separate cohort of participants than the main study (recruitment started on 14 July 2025). Data for the addendum arms will not be reported for Primary Outcome Measures. Participant Flow, Baseline Characteristics, and Adverse Events data for the addendum arms will be reported at the time of final results reporting.
Period: Overall Study
Arm/Group | 1400 mg Donanemab - Standard Regimen | 1400 mg Donanemab - Dose Skipping | 1400 mg Donanemab - Titration | 1400 mg Donanemab - Maximum Concentration (Cmax)
Started | 208 | 210 | 212 | 213
Received At Least 1 Dose of Study Drug | 207 | 210 | 212 | 213
Completed | 0 | 0 | 0 | 0
Not Completed | 208 | 210 | 212 | 213
Not completed — Continuing Study | 194 | 196 | 193 | 191
Not completed — Withdrawal by Subject | 8 | 5 | 7 | 13
Not completed — Adverse Event | 4 | 6 | 4 | 5
Not completed — Physician Decision | 0 | 2 | 4 | 1
Not completed — Lost to Follow-up | 1 | 1 | 2 | 1
Not completed — Participant was Non-ambulatory | 0 | 0 | 1 | 0
Not completed — Participant had Poor Venous Access | 0 | 0 | 0 | 1
Not completed — Assigned Treatment by Mistake | 0 | 0 | 0 | 1
Not completed — Death | 0 | 0 | 1 | 0
Not completed — Withdrawal Due to Caregiver Circumstances | 1 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Population: All participants who received at least one dose of donanemab.
Groups:
- 1400 mg Donanemab - Standard Regimen: Participants received:
  * 700 mg donanemab administered IV at baseline, week 4, and 8.
  * placebo administered IV at week 2, 6, 10, and 14.
  * 1400 mg of donanemab administered IV at week 12, 16, 20, and 24.
- 1400 mg Donanemab - Cmax: Participants received:
  * 350 mg donanemab administered IV at baseline, weeks 2, 4, 6, 8, and 10.
  * 700 mg donanemab administered IV at weeks 12 and 14.
  * 1400 mg of donanemab administered IV at weeks 16, 20, and 24.
- Total: Total of all reporting groups
Arm/Group | 1400 mg Donanemab - Standard Regimen | 1400 mg Donanemab - Dose Skipping | 1400 mg Donanemab - Titration | 1400 mg Donanemab - Cmax | Total
Number analyzed (Participants) | 207 | 210 | 212 | 213 | 842
Age, Continuous [Mean (Standard Deviation); unit: years] | 73.30 (5.66) | 73.40 (5.80) | 74.30 (5.69) | 73.20 (6.02) | 73.60 (5.80)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 120 | 117 | 126 | 123 | 486
  Male | 87 | 93 | 86 | 90 | 356
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 11 | 9 | 11 | 15 | 46
  Not Hispanic or Latino | 189 | 193 | 195 | 190 | 767
  Unknown or Not Reported | 7 | 8 | 6 | 8 | 29
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 1 | 0 | 0 | 1
  Asian | 0 | 3 | 3 | 3 | 9
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 0
  Black or African American | 11 | 8 | 14 | 13 | 46
  White | 196 | 197 | 193 | 196 | 782
  More than one race | 0 | 1 | 2 | 1 | 4
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0
Region of Enrollment [Count of Participants; unit: Participants]
  United Kingdom | 20 | 28 | 20 | 27 | 95
  United States | 187 | 182 | 192 | 186 | 747

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants With Any Occurrence of Amyloid-Related Imaging Abnormality-Edema/Effusion (ARIA-E)
Description: Percentage of participants with occurrence of ARIA-E at Week 24 is reported here.
Time Frame: 24 Weeks
Population: All participants who received at least one dose of donanemab and had evaluable data for this outcome.
Measure: Number; unit: Percentage of participants
Arm/Group | 1400 mg Donanemab - Standard Regimen | 1400 mg Donanemab - Dose Skipping | 1400 mg Donanemab - Titration | 1400 mg Donanemab - Cmax
Number analyzed (Participants) | 207 | 210 | 212 | 213
Percentage of participants | 23.67 | 18.57 | 13.68 | 18.31

2. Secondary Outcome: Percentage of Participants With Any Occurrence of ARIA-E
Description: Outcome data will be provided after the study is completed.
Time Frame: 52 Weeks
Reporting Status: Not Posted, anticipated posting 2026-05

3. Secondary Outcome: Change From Baseline in Brain Amyloid Plaque Deposition As Measured By Amyloid Positron Emission Tomography (PET) Scan
Description: Outcome data will be provided after the study is completed.
Time Frame: Baseline, 76 Weeks
Reporting Status: Not Posted, anticipated posting 2026-05

4. Secondary Outcome: Percentage of Participants With Any Occurrence of Amyloid-Related Imaging Abnormality-Hemorrhage/Hemosiderin Deposits (ARIA-H)
Description: Percentage of participants with occurrence of ARIA-H at Week 24 is reported here.
Time Frame: 24 Weeks
Population: All participants who received at least one dose of donanemab and had evaluable data for this outcome.
Measure: Number; unit: Percentage of participants
Arm/Group | 1400 mg Donanemab - Standard Regimen | 1400 mg Donanemab - Dose Skipping | 1400 mg Donanemab - Titration | 1400 mg Donanemab - Cmax
Number analyzed (Participants) | 207 | 210 | 212 | 213
Percentage of participants | 25.12 | 22.86 | 20.28 | 20.66

5. Secondary Outcome: Percentage of Participants With ARIA-H
Description: Outcome data will be provided after the study is completed.
Time Frame: 52 Weeks
Reporting Status: Not Posted, anticipated posting 2026-05

6. Secondary Outcome: Percentage of Participants With Maximum Severity of ARIA-E or ARIA-H
Description: Outcome data will be provided after the study is completed.
Time Frame: 76 Weeks
Reporting Status: Not Posted, anticipated posting 2026-05

7. Secondary Outcome: Pharmacokinetics (PK): Average Serum Concentration of Donanemab
Description: Outcome data will be provided after the study is completed.
Time Frame: Baseline to 76 Weeks
Reporting Status: Not Posted, anticipated posting 2026-05

8. Secondary Outcome: Number of Participants With Anti-Drug Antibodies (ADAs) Against Donanemab, Including Treatment Emergent ADAs and Neutralizing Antibodies
Description: Outcome data will be provided after the study is completed.
Time Frame: Baseline to End of Follow-Up (91 Weeks)
Reporting Status: Not Posted, anticipated posting 2026-05

ADVERSE EVENTS:
Time Frame: Baseline Up To 24 Weeks
Description: All participants who received at least one dose of donanemab. As pre-specified in statistical analysis plan, adverse events were reported per treatment arms.
Groups:
- 1400 mg Donanemab - Standard Regimen: Participants received:
  * 700 mg donanemab administered IV at baseline, week 4, and 8. placebo administered IV at week 2, 6, 10, and 14.
  * 1400 mg of donanemab administered IV at week 12, 16, 20, and 24.
Arm/Group | 1400 mg Donanemab - Standard Regimen | 1400 mg Donanemab - Dose Skipping | 1400 mg Donanemab - Titration | 1400 mg Donanemab - Cmax
All-Cause Mortality (participants affected / at risk) | 0/207 | 0/210 | 1/212 | 0/213
Serious Adverse Events (participants affected / at risk) | 18/207 | 18/210 | 23/212 | 20/213
Other Adverse Events (participants affected / at risk) | 139/207 | 140/210 | 141/212 | 137/213
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | 1400 mg Donanemab - Standard Regimen (N=207) | 1400 mg Donanemab - Dose Skipping (N=210) | 1400 mg Donanemab - Titration (N=212) | 1400 mg Donanemab - Cmax (N=213)
Atrial fibrillation (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Bradycardia (Cardiac disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Cardiac failure congestive (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Coronary artery disease (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Myocardial infarction (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Colitis (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Duodenal ulcer (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Gastric haemorrhage (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Gastrointestinal haemorrhage (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Incarcerated inguinal hernia (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Large intestine perforation (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Pancreatitis acute (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Small intestinal obstruction (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Upper gastrointestinal haemorrhage (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Vomiting (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Chest pain (General disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Cholelithiasis (Hepatobiliary disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Anaphylactic reaction (Immune system disorders) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Drug hypersensitivity (Immune system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Arthritis infective (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Bronchitis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Cellulitis (Infections and infestations) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Clostridium difficile infection (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Diverticulitis (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Laryngitis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Osteomyelitis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Pneumonia (Infections and infestations) | 1 (1) | 1 (1) | 1 (2) | 0 (0)
Respiratory syncytial virus infection (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Sepsis (Infections and infestations) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
Urosepsis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Cervical vertebral fracture (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Fall (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Femur fracture (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Fractured coccyx (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Hip fracture (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 2 (2) | 1 (1)
Infusion related reaction (Injury, poisoning and procedural complications) | 1 (1) | 1 (1) | 2 (2) | 2 (2)
Pelvic fracture (Injury, poisoning and procedural complications) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Procedural pain (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Road traffic accident (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Hypokalaemia (Metabolism and nutrition disorders) | 0 (0) | 2 (2) | 0 (0) | 0 (0)
Hyponatraemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Lactic acidosis (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Malnutrition (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Compartment syndrome (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (3) | 0 (0)
Chronic lymphocytic leukaemia (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Clear cell renal cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Follicular lymphoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Amyloid related imaging abnormality-oedema/effusion (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Cerebral haemorrhage (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Cerebral infarction (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Cerebral venous sinus thrombosis (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Cerebrovascular accident (Nervous system disorders) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
Headache (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Hemiparesis (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Ischaemic stroke (Nervous system disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Metabolic encephalopathy (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Middle cerebral artery stroke (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Myelopathy (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Seizure (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Syncope (Nervous system disorders) | 2 (4) | 0 (0) | 2 (2) | 1 (1)
Transient ischaemic attack (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Mental status changes (Psychiatric disorders) | 1 (2) | 0 (0) | 0 (0) | 0 (0)
Suicidal ideation (Psychiatric disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Acute respiratory failure (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
Asthma (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Cough (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Tracheomalacia (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Aortic stenosis (Vascular disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Axillary vein thrombosis (Vascular disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Haematoma (Vascular disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Hypertension (Vascular disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Hypertensive crisis (Vascular disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Hypotension (Vascular disorders) | 0 (0) | 1 (1) | 1 (1) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | 1400 mg Donanemab - Standard Regimen (N=207) | 1400 mg Donanemab - Dose Skipping (N=210) | 1400 mg Donanemab - Titration (N=212) | 1400 mg Donanemab - Cmax (N=213)
Diarrhoea (Gastrointestinal disorders) | 12 (15) | 12 (12) | 6 (8) | 15 (15)
Fatigue (General disorders) | 11 (19) | 8 (8) | 12 (14) | 11 (12)
Covid-19 (Infections and infestations) | 10 (10) | 16 (16) | 19 (19) | 12 (12)
Upper respiratory tract infection (Infections and infestations) | 8 (9) | 14 (14) | 8 (8) | 7 (8)
Urinary tract infection (Infections and infestations) | 7 (7) | 18 (23) | 16 (19) | 9 (9)
Fall (Injury, poisoning and procedural complications) | 16 (26) | 17 (21) | 19 (20) | 19 (23)
Infusion related reaction (Injury, poisoning and procedural complications) | 27 (42) | 18 (27) | 34 (69) | 41 (86)
Arthralgia (Musculoskeletal and connective tissue disorders) | 8 (9) | 5 (6) | 13 (14) | 4 (5)
Amyloid related imaging abnormality-microhaemorrhages and haemosiderin deposits (Nervous system disorders) | 33 (38) | 33 (40) | 28 (32) | 37 (47)
Amyloid related imaging abnormality-oedema/effusion (Nervous system disorders) | 49 (58) | 38 (40) | 29 (32) | 39 (41)
Dizziness (Nervous system disorders) | 19 (20) | 16 (18) | 17 (17) | 10 (13)
Headache (Nervous system disorders) | 41 (88) | 44 (54) | 32 (42) | 33 (37)
Superficial siderosis of central nervous system (Nervous system disorders) | 12 (14) | 13 (20) | 5 (6) | 4 (4)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of more than 60 days

DOCUMENTS (2):
  • Study Protocol (2023-05-26): https://cdn.clinicaltrials.gov/large-docs/86/NCT05738486/Prot_000.pdf
  • Statistical Analysis Plan (2024-07-29): https://cdn.clinicaltrials.gov/large-docs/86/NCT05738486/SAP_001.pdf